CLINICAL TRIAL: NCT06364163
Title: A Study on the Effect of Consuming a Herring Oil Concentrate on LDL Cholesterol Concentration in Adults With Overweight or Obesity
Brief Title: Effect of Herring Oil Concentrate on LDL Cholesterol Concentration in Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Norwegian Seafood Research Fund (Unknown)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 697716
Record Dates: First submitted 2024-04-06; First posted 2024-04-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: High Cholesterol
Keywords: Cholesterol; Cetoleic acid
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herring oil concentrate (Experimental): Dietary supplement: herring oil concentrate in capsules, 4 g oil daily for 8 weeks
  Interventions: Dietary Supplement: Herring oil concentrate
- Control oil (Placebo Comparator): Dietary supplement: control oil in capsules, 4 g oil daily for 8 weeks
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Herring oil concentrate — Capsules containing herring oil concentrate, taken daily for 8 weeks.
  Arms: Herring oil concentrate
Dietary Supplement: Control — Capsules containing control oil, taken daily for 8 weeks.
  Arms: Control oil

SUMMARY:
High cholesterol concentration is a major risk factor for cardiovascular disease (CVD), and consumption of fish has been associated with a lower CVD risk in several studies. The beneficial health effects of consuming fish have traditionally been ascribed to the long-chain PUFA (LC-PUFA) EPA (C20:5n-3) and DHA (C22:6n-3), although consumption of fish oils or concentrates with high EPA and DHA contents does not affect the cholesterol concentration in humans and lowers the cholesterol concentration in rats and mice only when given in very high doses. Fish oils contain a plethora of fatty acids besides EPA and DHA, and in recent years, increased focus has been on the long-chain MUFA (LC-MUFA) cetoleic acid (C22:1n-11). Cetoleic acid is found in high amounts in oils from certain fish species such as herring, which has relatively low contents of both EPA and DHA. The investigators have recently summarised and meta-analysed the available literature that investigates the effects of diets containing fish oils or fish oil concentrates that have a high content of cetoleic acid but low or no content of EPA and DHA on cholesterol concentration in rodents, showing that cetoleic acid-rich fish oils and concentrates prevent high cholesterol concentration.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 25 kg/m2
* Stable body weight last 3 months

Exclusion Criteria:

* Allergies towards fish, milk, egg, gluten
* Tobacco use (cigarettes or snus)
* Diseases affecting the heart, intestinal function, kidney function or insulin secretion
* Use of medications targeting cholesterol -or glucose metabolism
* Use of dietary supplements
* Pregnant or breastfeeding
* Following a strict diet
* Had bariatric surgery or using medications for weight loss
* Recent or planned surgical procedures
* High intake of fish/seafood

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of LDL-cholesterol | 8 weeks
  LDL-cholesterol will be measured in fasting serum samples

SECONDARY OUTCOMES:
Serum concentration of HDL-cholesterol | 8 weeks
  HDL-cholesterol will be measured in fasting serum samples
Serum concentration of total cholesterol | 8 weeks
  Total cholesterol will be measured in fasting serum samples
Serum concentrations of apolipoproteins | 8 weeks
  Lipoproteins will be measured in fasting serum samples
Serum concentrations of amino acids metabolites | 8 weeks
  Metabolites of amino acids will be measured in fasting serum samples
Serum concentration of one-carbon pathway metabolites | 8 weeks
  Metabolites in the one-carbon pathway will be measured in fasting serum samples
Fatty acid composition in leukocytes | 8 weeks
  Leukocytes will be isolated from fasting serum before quantification of fatty acids
Serum concentration of glucose | 8 weeks
  Glucose will be measured in serum sampled in fasting condition
Serum concentration of insulin | 8 weeks
  Insulin will be measured in serum sampled in fasting condition
Body composition | 8 weeks
  Percent body fat will be measured using bioimpedance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No